CLINICAL TRIAL: NCT04010058
Title: Postoperative Continuous Non-invasive Haemodynamic Monitoring on the Ward: a Feasibility Study
Brief Title: Postoperative Continuous Non-invasive Haemodynamic Monitoring on the Ward
Acronym: PostConMon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19SURN268889
Record Dates: First submitted 2019-06-27; First posted 2019-07-08 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Surgical Procedures, Operative; Hemodynamic Instability; Blood Pressure Disorders

STUDY DESIGN:
Intervention Model Description: This is a feasibility study of the use of an approved device (CE-marked) in a cohort of postoperative patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LIDCO CNAP device — The LiDCO CNAP device (referred to as CNAP in this document) provides continuous cardiac output non-invasively, without the requirement for an arterial catheter. It uses a dual finger cuff in addition to a standard arm cuff (familiar to everyone who's had their blood pressure checked) and it transforms infrared plethysmographic signals into continuous blood pressure information. It uses an algorithm to derive cardiac output-related parameters. In recognition of the potential difference between the derived values and any measured values, it refers to some of its values as 'nominal' values. It has been evaluated in a range of surgical populations8-11 a post-operative cohort12, and a haemodynamically unstable critical care population13. In a population of patients undergoing endoscopy there was increased detection of episodes of hypotension compared with standard measures.

SUMMARY:
The patient's clinical care will not be altered apart from an the use of a non-invasive monitor for a short time, without any biological sample acquisition, or follow-up. This is low risk.

The device works through a complex pressure measurement in the fingers and by slightly squashing the fingers it can cause minor impairments to circulation. This represents a very small risk. To mitigate this risk the investigators will exclude patients with impaired circulation to the fingers and fingers will be monitored.

The approach is necessarily on the day of surgery and for many people this is an anxious time. The investigators have a lot of experience of approaching patients on the day of surgery for providing consent for observational studies - the investigators use caution and sensitivity. The investigators do not approach patients who the clinical team consider anxious or where there is significant pressure on time.

DETAILED DESCRIPTION:
Enrolled patients will have the CNAP sited in the post-anaesthetic care unit (PACU) and it will stay on their arm until at least 12 hours have passed. The device will collect continuous heart rate, blood pressure, and nominal cardiac output; it also derives a range of values from these measurements. There is minimal risk attributable to the use of the CNAP device. These devices are already in routine clinical use in the UK in intensive care units, high-dependency units and operating theatres.

To reduce burden on the patient, no additional HR/BP monitor is required and whenever the usual care team would like to know the HR or BP these values will be displayed. The additional parameters (related to measurement of cardiac output) will not be shared with the clinical team - they will remain blinded to these data because otherwise there is the risk that they would use this additional information to alter clinical management.

Medical notes will be examined to provide information about demographics, physical characteristics (height, weight), and previous medical history - please see case report form (CRF, appendix 1) for more details.

There are no blood tests, or other acquisition of biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Has capacity to provide informed consent
* Surgery: planned or unplanned; all types including gastrointestinal, urology, orthopaedics and gynaecological
* Due for an inpatient stay (i.e. not day case surgery) on either Frensham or Bramshott wards (staff will have had training with the device on these wards)
* Aged 18 years or over

Exclusion Criteria:

* Admission to intensive care unit ICU / high dependency unit HDU
* Declines consent to participate, or lack capacity to provide consent
* Impaired circulation of the hands: Raynaud's disease or severe peripheral vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2019-11-22 (Estimated); Study Completion 2019-11-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 3 months
  Number of suitable patients who provide consent and have the device sited / number of suitable patients who provide consent (%)
Acceptability | 3 months
  In those patients who have provided consent and had the monitor sited, how many tolerate the device and keep it on throughout the observation period (at least 12 hours) and provide useable data / number of suitable patients who provide consent and have the device sited (%)

SECONDARY OUTCOMES:
What proportion of patients have any recorded episodes of hypotension? | 3 months
  Endpoint: proportion of patients with hypotension Outcome 1: number of patients with SBP<90mmHg / total number of patients (%)
What proportion of patients have any recorded episodes of hypotension? Just considering the time on the ward, after PACU | 3 months
  Endpoint: proportion of patients with hypotension Outcome: number of patients with SBP<90mmHg / total number of patients (%)
In the PACU, considering those with at least one episode of SBP<90mmHg, how long are patients hypotensive for? (CNAP data) | 3 months
  Endpoint: duration of hypotension, sum of all episodes Outcome 1: minutes of hypotension Outcome 2: proportion of total time in PACU with hypotension
On the ward, considering those with at least one episode of SBP<90mmHg, when using data from the CNAP, how long are patients hypotensive for? | 3 months
  Duration of hypotension from CNAP, sum of all episodes (CNAP min) Episodes of hypotension with CNAP, total duration as sum of individual episode durations
On the ward, considering those with at least one episode of SBP<90mmHg, when using data from VitalPAC, how long are patients hypotensive for? | 3 months
  Duration of hypotension from VitalPAC, sum of all episodes (VitalPACmin) Episodes of hypotension with VitalPAC, total duration as sum of individual episode durations
On the ward, when there are discrete episodes of hypotension, what is the distribution of nominal stroke volume index? | 3 months
  nominal stroke volume index (nSVI) Outcome 1: Histogram of nSVI Outcome 2: Proportion of episodes of hypotension with an nSVI: low (<35ml/m2), normal (35-65ml/m2) and high (>65ml/m2)
On the ward, when there are discrete episodes of hypotension, when paired with MAP and a notional RAP, what is the distribution of systemic vascular resistance index, SVRI? | 3 months
  systemic vascular resistance index (SVRI) Distribution of SVRI
During an episode of hypotension, what intravenous fluids are given, at what prescribed rate? | 3 months
  Endpoint: observation of clinical care Outcome: which intravenous fluids, at what prescribed rate?
During episodes of hypotension treated with an intravenous fluid bolus (IVFB) what is the haemodynamic response? Is the response predictable using either baseline nSVI or SVV? | 3 months
  Endpoint: SBP and nSVI before and during/after IVFB (30 minutes after start) Outcome 1: Categorise episodes into the following: responders (≥15% increase in nSVI or ≥15% SBP) or non-responders (<15% increase in nSVI and SBP) Outcome 2: Display distribution of nSVI (low/normal/high) prior to IVFB between responders and non-responders.
  Outcome 3: Compare % change in nSVI in response to IVFB between those with low nSVI (potentially more responsive) to normal/high nSVI.
  Outcome 4: Compare SVV (%) measured before IVFB between responders and non-responders.
What proportion of IVF boluses are associated with a significant improvement in haemodynamics? | 3 months
  Endpoint: Number of IVFB that are associated with haemodynamic benefit (≥15% increase in nSVI or ≥15% SBP) / Total number of IVFB
Volume of IVF given that would not have been indicated by CNAP readings | 3 months
  Endpoint: Sum of individual IVF boluses given when both of the following conditions are met at the start of the IVF bolus:
  1. Prior IVF did not improve nSVI by ≥15%
  2. Stroke Volume Variation <5%
What treatments were delivered intra-operatively and in PACU. | 3 months
  Endpoint: observation of clinical care Outcome: Receipt of intravenous fluids, blood products, vasopressor drugs, admission to critical care.
What are the clinical outcomes? length of stay (LOS) | 3 months
  Clinical outcomes from medical records : length of stay (LOS)
What are the clinical outcomes? critical care admission | 3 months
  Endpoint: Clinical outcomes from medical records: critical care admission (ICU LOS)
What are the clinical outcomes? acute kidney injury | 3 months
  Endpoint: Clinical outcomes from medical records: acute kidney injury (from urine output and change in creatinine)
What are the clinical outcomes? acute myocardial infarction | 3 months
  Endpoint: Clinical outcomes from medical records: acute myocardial infarction (EPCO definition)
What are the clinical outcomes? incidence of blood transfusion | 3 months
  Endpoint: Clinical outcomes from medical records: incidence of blood transfusion
What are the clinical outcomes? unplanned ICU admission | 3 months
  Endpoint: Clinical outcomes from medical records: unplanned ICU admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey County Hospital, Guildford, United Kingdom

REFERENCES:
- [Derived] King CE, Kermode A, Saxena G, Carvelli P, Edwards M, Creagh-Brown BC. Postoperative continuous non-invasive cardiac output monitoring on the ward: a feasibility study. J Clin Monit Comput. 2021 Dec;35(6):1349-1356. doi: 10.1007/s10877-020-00601-z. Epub 2020 Oct 22. PMID 33094826